CLINICAL TRIAL: NCT00188149
Title: Optimization of the Primary Therapy for Patients With Hodgkin's Lymphoma and Evaluation of the Positron Emission Tomography (PET) as a Diagnostic Tool for Primary Staging and Assessment of the Effects of the Therapy
Brief Title: Optimization of the Primary Therapy for Patients With Hodgkin's Disease and Evaluation of PET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Carl Gustav Carus (Other)
Collaborators: Technische Universität Dresden (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGC05MK1002
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2005-09

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin's Lymphoma; Chemotherapy; Radiation therapy; PET
MeSH Terms: conditions — Hodgkin Disease | interventions — ABVD protocol; Radiotherapy

INTERVENTIONS:
Drug: Combined chemotherapy (ABVD, BACOPP-D)
Procedure: Radiation therapy

SUMMARY:
Prognosis of patients with Hodgkin´s lymphoma (HL) has been improved significantly over the last decade. Therefore, the impact of treatment associated long-term toxicities and late effects such as second cancers increased. The purpose of this prospective multicenter trial is to show the feasibility of the treatment with ABVD alone in patients with limited stage (HL1) and intermediate stage (HL2) disease and of an intensified etoposide-free chemotherapy regimen for patients with advanced disease (HL3) including 18F-FDG-PET evaluation.

DETAILED DESCRIPTION:
The aim in limited and intermediate stages is to reduce the toxicity by omitting the subsequent radiotherapy in patients with complete remission after ABVD chemotherapy. Patients with limited disease receive four cycles, patients with intermediate disease (according to the criteria of the German Hodgkin Study group, GHSG) receice six cycles of ABVD. In case of residual mass (> 1.5 cm), additional involved field irradiation is planned. The aim in advanced disease using BACOPP-D regimen which includes cyclophosphamide, adriamycin, dacarbazine, procarbazine, prednisolone, bleomycin and vincristine, is to reduce the hematological toxicity and the secondary leukemias by omitting etoposide (in comparison to the BEACOPP escalated regimen). All patients receive eight cycles of the BACOPP-D regimen. In case of residual mass (> 1.5 cm), additional involved field irradiation is planned. Additionally, we want to evaluate the CT- and PET-based remission status after chemotherapy and at final staging.

ELIGIBILITY:
Inclusion Criteria (HL1):

* Histologically confirmed Hodgkin´s Lymphoma (WHO Classification 1999)

  1. Classical Hodgkin Lymphoma: Nodular sclerosis (type 1 and 2) / Mixed type / Lymphocyte depleted type / Lymphocyte rich type
  2. Nodular lymphocyte-predominant Hodgkin Lymphoma
* Patients in stage: Clinical stage (CS) I without risk factors / CS II without risk factors
* Age between 16 and 75
* Written informed consent

Inclusion criteria (HL2):

* Histologically confirmed Hodgkin´s Lymphoma (WHO Classification 1999)

  1. Classical Hodgkin´s Lymphoma: Nodular sclerosis (type 1 and 2) / Mixed type / Lymphocyte depleted type / Lymphocyte rich type
  2. Nodular lymphocyte-predominant Hodgkin Lymphoma
* Patients in stage

  1. Clinical stage (CS) I,II A with risk factors: Large mediastinal tumor (>1/3 of the maximal diameter of the thoracic cavity) / Extranodal disease / Sedimentation rate ≥ 50 mm/h for patients without B-symptomes or ≥ 30 mm/h for patients with B-symptomes / ≥ 3 lymph node areas infiltrated with tumor cells
  2. Clinical stage (CS) II B with risk factors: Sedimentation rate ≥ 50 mm/h for patients without B-symptomes or ≥ 30 mm/h for patients with B-symptomes / ≥ 3 lymph node areas infiltrated with tumor cells
* Age between 16 and 75
* Written informed consent

Inclusion criteria (HL3):

* Histologically confirmed Hodgkin´s Lymphoma (WHO Classification 1999)

  1. Classical Hodgkin's Lymphoma (Hodgkin's desease): Nodular sclerosis (type 1 and 2) / Mixed type / Lymphocyte depleted type / Lymphocyte rich type
  2. Nodular lymphocyte-predominant Hodgkin Lymphoma
* Patients in stage

  1. Clinical stage (CS) II B with minimum one of the following risk factors: Large mediastinal tumor (≥1/3 of the maximal diameter of the thoracic cavity) / Extranodal disease
  2. Clinical stage (CS) III
  3. Clinical stage (CS) IV
* Age between 16 and 65
* Written informed consent

Exclusion Criteria (HL1, HL2 and HL3):

* Poor general condition not related to the lymphoma (ECOG perfomance status 3 or 4; Karnofsky Index < 50 %)
* Severe concomitant diseases: cardiac insufficiency (NYHA grade III or IV) / chronic respiratory insufficiency with hypoxemia / Hepatic insufficiency (cirrhosis, Hepatitis B or C / chronic renal insufficiency / HIV infection or other out-of-control infections / hematopoetic insufficiency (Leukocytes < 3000/µl; Thrombocytes < 100.000/µl / psychiatric diseases
* History of previous malignancy in the last 5 years
* Pregnancy
* Patients not likely to comply to the requirements stemming form the participation in the trial

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2000-05; Study Completion 2007-12

PRIMARY OUTCOMES:
- Feasibility and acute toxicity of the therapy
- The Free from Therapy Failure (FFTF) rate after one year
- Event-Free Survival (EFS) rate and overall survival rate
- Evaluation of the PET as a diagnostic tool for the primary tumor staging as well for assessment of the effects of the therapy

SECONDARY OUTCOMES:
- Evaluation of the quality of life of the patients during and after the therapy
- Occurence of late toxicity after the end of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Naumann, MD, Principal Investigator — University Clinic "Carl Gustav Carus" Dresden
Locations (1):
- Medizinische Klinik und Poliklinik I, University Clinic Carl Gustav Carus, Dresden, Saxony, Germany

REFERENCES:
- [Background] Anselmo AP, Bove M, Cartoni C, Damico C, Maurizi Enrici R, Falchetto Osti M, Biagini C. Combined modality (ABVD plus radiotherapy) versus radiotherapy in the management of early stage (IIA) Hodgkin's disease with mediastinal involvement. Haematologica. 1992 Mar-Apr;77(2):177-9. PMID 1383107
- [Background] Biti GP, Cimino G, Cartoni C, Magrini SM, Anselmo AP, Enrici RM, Bellesi GP, Bosi A, Papa G, Giannarelli D, et al. Extended-field radiotherapy is superior to MOPP chemotherapy for the treatment of pathologic stage I-IIA Hodgkin's disease: eight-year update of an Italian prospective randomized study. J Clin Oncol. 1992 Mar;10(3):378-82. doi: 10.1200/JCO.1992.10.3.378. PMID 1740677
- [Background] Canellos GP, Anderson JR, Propert KJ, Nissen N, Cooper MR, Henderson ES, Green MR, Gottlieb A, Peterson BA. Chemotherapy of advanced Hodgkin's disease with MOPP, ABVD, or MOPP alternating with ABVD. N Engl J Med. 1992 Nov 19;327(21):1478-84. doi: 10.1056/NEJM199211193272102. PMID 1383821
- [Background] Carde P, Hagenbeek A, Hayat M, Monconduit M, Thomas J, Burgers MJ, Noordijk EM, Tanguy A, Meerwaldt JH, Le Fur R, et al. Clinical staging versus laparotomy and combined modality with MOPP versus ABVD in early-stage Hodgkin's disease: the H6 twin randomized trials from the European Organization for Research and Treatment of Cancer Lymphoma Cooperative Group. J Clin Oncol. 1993 Nov;11(11):2258-72. doi: 10.1200/JCO.1993.11.11.2258. PMID 7693881
- [Background] Cosset JM, Henry-Amar M, Meerwaldt JH, Carde P, Noordijk EM, Thomas J, Burgers JM, Somers R, Hayat M, Tubiana M. The EORTC trials for limited stage Hodgkin's disease. The EORTC Lymphoma Cooperative Group. Eur J Cancer. 1992;28A(11):1847-50. doi: 10.1016/0959-8049(92)90018-w. No abstract available. PMID 1389523
- [Background] Diehl V, Sieber M, Ruffer U, Lathan B, Hasenclever D, Pfreundschuh M, Loeffler M, Lieberz D, Koch P, Adler M, Tesch H. BEACOPP: an intensified chemotherapy regimen in advanced Hodgkin's disease. The German Hodgkin's Lymphoma Study Group. Ann Oncol. 1997 Feb;8(2):143-8. doi: 10.1023/a:1008294312741. PMID 9093722
- [Background] Fleming TR. One-sample multiple testing procedure for phase II clinical trials. Biometrics. 1982 Mar;38(1):143-51. PMID 7082756
- [Background] GEHAN EA. A GENERALIZED WILCOXON TEST FOR COMPARING ARBITRARILY SINGLY-CENSORED SAMPLES. Biometrika. 1965 Jun;52:203-23. No abstract available. PMID 14341275
- [Background] Horning SJ, Hoppe RT, Mason J, Brown BW, Hancock SL, Baer D, Rosenberg SA. Stanford-Kaiser Permanente G1 study for clinical stage I to IIA Hodgkin's disease: subtotal lymphoid irradiation versus vinblastine, methotrexate, and bleomycin chemotherapy and regional irradiation. J Clin Oncol. 1997 May;15(5):1736-44. doi: 10.1200/JCO.1997.15.5.1736. PMID 9164180
- [Background] Longo DL, Glatstein E, Duffey PL, Young RC, Hubbard SM, Urba WJ, Wesley MN, Raubitschek A, Jaffe ES, Wiernik PH, et al. Radiation therapy versus combination chemotherapy in the treatment of early-stage Hodgkin's disease: seven-year results of a prospective randomized trial. J Clin Oncol. 1991 Jun;9(6):906-17. doi: 10.1200/JCO.1991.9.6.906. PMID 2033427
- [Background] Peto R, Pike MC, Armitage P, Breslow NE, Cox DR, Howard SV, Mantel N, McPherson K, Peto J, Smith PG. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. II. analysis and examples. Br J Cancer. 1977 Jan;35(1):1-39. doi: 10.1038/bjc.1977.1. PMID 831755
- [Background] Ruiz-Arguelles GJ, Gomez-Almaguer D, Apreza-Molina MG. Chemotherapy alone may be an efficient alternative in the treatment of early stage Hodgkin's disease if optimal radiotherapy is not available. Leuk Lymphoma. 1997 Sep;27(1-2):179-83. doi: 10.3109/10428199709068285. PMID 9373210
- [Background] Salloum E, Doria R, Schubert W, Zelterman D, Holford T, Roberts KB, Farber LR, Kiehl RK, Cardinale J, Cooper DL. Second solid tumors in patients with Hodgkin's disease cured after radiation or chemotherapy plus adjuvant low-dose radiation. J Clin Oncol. 1996 Sep;14(9):2435-43. doi: 10.1200/JCO.1996.14.9.2435. PMID 8823321
- [Background] Seegenschmiedt MH. Interdisciplinary documentation of treatment side effects in oncology. Present status and perspectives. Strahlenther Onkol. 1998 Nov;174 Suppl 3:25-9. PMID 9830452
- [Background] Specht L, Gray RG, Clarke MJ, Peto R. Influence of more extensive radiotherapy and adjuvant chemotherapy on long-term outcome of early-stage Hodgkin's disease: a meta-analysis of 23 randomized trials involving 3,888 patients. International Hodgkin's Disease Collaborative Group. J Clin Oncol. 1998 Mar;16(3):830-43. doi: 10.1200/JCO.1998.16.3.830. PMID 9508163
- [Background] Wirth A, Corry J, Laidlaw C, Matthews J, Liew KH. Salvage radiotherapy for Hodgkin's disease following chemotherapy failure. Int J Radiat Oncol Biol Phys. 1997 Oct 1;39(3):599-607. doi: 10.1016/s0360-3016(97)00352-0. PMID 9336139